CLINICAL TRIAL: NCT06548334
Title: The Effectiveness of Lumber Regression Technique on Disc Bulge Randomized Control Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/736
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Disc Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced Physiotherapy (Experimental)
  Interventions: Combination Product: Advanced Physiotherapy
- Conventional Physiotherapytechniques (Active Comparator)
  Interventions: Other: Conventional Physiotherapy Techniques

INTERVENTIONS:
Combination Product: Advanced Physiotherapy — The physiotherapist used the regression techniques for 1 hour of session 2 times for 8 weeks. The caudal component involved the spinous process of the treated segment touching the therapist's hand and not applying force as though mobilising the segment at grade 2. These were applied if there is a suspected case of a posterolateral disc prolapse where the aim is to increase the diameter of the foramen and decrease the tension exerted on the nerve root. Applied posteroanterior was used to distract the anterior intervertebral end plate and to approximate the posterior end plates so as to pull back the protruded nuclear material by creating a negative pressure.
  Arms: Advanced Physiotherapy
Other: Conventional Physiotherapy Techniques — In traditional physiotherapy, the patient underwent two sessions per week for eight weeks. Each session lasted one hour and included 20minutes of TENS treatment. The flexibility exercises consisted of hamstring stretches and single and double knee-to-chest stretches. The strengthening exercises were partial sit-ups, quadruped lifts, and double leg hold; pelvic tilts were performed with 10-15 repetitions, each held for 20-30 seconds and repeated three times.
  Arms: Conventional Physiotherapytechniques

SUMMARY:
Lumbar disc bulges lead to considerable pain and disability in affected individuals, with current interventions lacking consistency of outcomes. The lumbar regression method offered a hopeful, noninvasive option.

DETAILED DESCRIPTION:
this study was proposed to evaluate its efficacy in improving accessary lower limb flexibility and reducing functional disability and pain management. To provide evidence about its effectiveness and help with clinical practice, this study aimed to improve patient outcomes in subjects having lumbar disc bulges.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a diagnosis of Disc bulge confirmed by MRI.
* Between 18 and 65 years of age.
* Chronic low back pain from the last 3 months
* A stable treatment environment that allows intervention.
* Ability to understand and follow course directions.
* Willingness to give informed consent

Exclusion Criteria:

* Spondylolisthesis
* Spondylosis
* Vertebral fracture
* Lack of ava
* Further research interventions.
* Unstable medical condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Roland Morris disability questionnaire | 12 Months
  The Roland-Morris low back pain and disability questionnaire (RMD) was utilised to evaluate the quality of life prior to and following the completion of the treatment. This questionnaire has demonstrated strong validity and reliability. The score is measured on a scale of 0 to 24, and percentage scores were calculated for each participant. Greater scores indicate a greater level of disabilities. Its sensitivity is 95%, and its specificity is 69%.
Straight Leg Raise | 12 months
  The normal angle for an SLR is from 0-35 degrees, which signifies the least amount of strain. Stretched from 35-70 degrees, sciatic nerve root stretching is achieved, and possible problems such as herniated disc or radiculopathy may be evidenced. 70- 90 degrees reflect highest normal flexibility: it may be related to hip joint pathology or some other conditions which are not a result of nerve injury. During both the first evaluation and the final therapy, the SLR was assessed using a digital inclinometer (clinometer) installed on a Techno Camon 20 Android phone. The digital inclinometer has been found to exhibit high levels of reliability and validity

CONTACTS AND LOCATIONS:
Locations (1):
- Nemat Hospital & Heart Center, Manga Mandi, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No